CLINICAL TRIAL: NCT05477719
Title: Study Evaluating the Effect of Compression Stockings at Constant Pressure for 28 Days on the Number of Apneas/Hypopneas Per Hour of Sleep (Index of Apneas/Hypopneas) in Patients With Syndrome Obstructive Sleep Apnea/Hypopnea as Compared to no Treatment
Brief Title: Effect of Compression Stockings on the Number of Apneas/Hypopneas Per Hour of Sleep in Patients With Syndrome Obstructive Sleep Apnea/Hypopnea as Compared to no Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sigvaris France (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2021-A00826-35
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Sleep Apnea Syndromes
Keywords: Obstructive sleep apnea; Fluid; Sedentary living; Compression stockings
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression stockings - No Compression (Experimental): The patient will wear specific compression stockings in the first phase, and no compression in the second phase of the study
  Interventions: Device: Wearing of specific compression stockings
- No Compression - Compression stockings (Experimental): The patient won't wear anything in the first phase, and specific compression stockings in the second phase of the study
  Interventions: Device: Wearing of specific compression stockings

INTERVENTIONS:
Device: Wearing of specific compression stockings — The patient will wear specific compression stockings prevent the accumulation of fluids during the day in the lower part of the body and thus limiting the nocturnal drainage effect from the lower part of the body to the upper part of the body

SUMMARY:
The sleep apnea-hypopnea syndrome is characterized by the occurrence, during sleep, of abnormally frequent episodes of interruption of ventilation (apnea), or significant reduction in ventilation (hypopnea).

The main symptoms of sleep apnea-hypopnea syndrome are daytime sleepiness (caused by the fragmentation and breakdown of sleep) and nocturnal snoring; possibly accompanied by the following symptoms: non-restorative sleep, difficulty concentrating, nocturia, cognitive disorders, libido disorders.

The consequences of sleep apnea-hypopnea syndrome are multiple for the patient both in the short term and in the long term.

The short-term manifestations are as follows: daytime sleepiness, reduced alertness, difficulty driving (risk of road accidents), difficulty performing tasks (risk of accidents at work), memory and concentration problems , learning difficulties (especially in children), mood disorders. In the end, there is an alteration in the quality of life of the patient.

Sleep apnea-hypopnea syndrome also has long-term consequences: a link between sleep apnea-hypopnea syndrome and cardiovascular morbidity and mortality has been explored by several cohort studies.

Nasal ventilation by continuous positive airway pressure is considered the reference treatment for sleep apnea-hypopnea syndrome. The use of nasal ventilation by continuous positive airway pressure, compared to no treatment, is not associated with a reduced risk of cardiovascular outcomes or death in patients with sleep apnea according to a recent meta-analysis.

Mandibular advancement devices are an alternative treatment for nasal ventilation by continuous positive airway pressure. The acceptability of its treatments, whether nasal ventilation by continuous positive airway pressure or mandibular advancement devices, is not very good and some patients do not start treatment or abandon it because of the constraints related to these treatments. There is therefore a need to find other treatments.

The overnight rostral fluid displacement from the legs, related to prolonged sitting can generate edema in the neck, more precisely in the upper airways, and therefore obstructive respiratory dysfunctions responsible for sleep apnea-hypopnea syndrome. Correlations between nocturnal fluid shifts and the number of apneas/hypopneas have been demonstrated Previous studies has shown a reduction in the apnea-hypopnea index by the daytime preventive wearing of medical compression, which can reduce the extent of leg edema and the displacement of nocturnal fluids.

The aim of the present study is to show that daytime wearing of medical compression developed specifically to optimize its effect in this indication for 28 days versus not wearing it reduces the number of apneas/hypopneas in patients with sleep apnea-hypopnea syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patient with moderate to severe sleep apnea-hypopnea syndrome confirmed by polysomnography dating less than 3 months with an index of apneas/hypopneas ≥ 15 apneas-hypopneas/h

  1. having been previously treated with nasal ventilation by continuous positive airway pressure and mandibular orthosis and having stopped treatment for at least 10 days, regardless of the duration of use of these two treatments
  2. or never treated for their sleep apnea-hypopnea syndrome satisfying the following 3 criteria

     1. having 1 or 2 of the following signs daytime sleepiness, severe and daily snoring, feelings of suffocation or suffocation during sleep, daytime fatigue, nocturia, morning headaches.
     2. absence of serious cardiovascular or respiratory comorbidity
     3. absence of severe daytime sleepiness and/or accidental risk that could lead to direct or indirect bodily harm
* stable weight (5% variation of the weight at the time of the polysomnography done within 3 months)
* patient without varicose veins, without trophic disorder that could suggest moderate to severe superficial or deep venous insufficiency (dermatitis, hypodermatitis, active or healed ulcer)
* sedentary patient (patient seated more than 8 h/d

Exclusion Criteria:

* daily wearing of medical compression
* patient with a contraindication to wearing a compression garment
* patient unable to apply compression (preliminary test)
* taking diuretics or venotonics
* obesity (body mass index > 30 kg/m2)
* patient with leg dermatosis
* patient with leg or thigh muscle trauma less than three months old
* patient with sciatica, cruralgia or acute low back pain
* pregnant or post-pregnancy women less than 6 months old or of childbearing age without an effective method of contraception
* heart, liver or kidney failure
* lymphedema of the lower limbs
* cancer not considered to be in remission
* history of abdominal radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the number of apneas/hypopneas | 28 days

SECONDARY OUTCOMES:
Proportion of patients with a 50% reduction in the apnea-hypopnea index | 28 days
Proportion of patients with an apnea-hypopnea index < 30/hour | 28 days
Proportion of patients with an apnea-hypopnea index < 15/hour | 28 days
Proportion of patients with a 50% reduction in the apnea-hypopnea index and an apnea-hypopnea index < 15/hour | 28 days
Change in sleep habits and characteristics | 28 days
  Change in sleep habits and characteristics will be evaluated with an ad hoc questionnaire
Change in sleepiness | 28 days
  Sleepiness will be assessed by Epworth scale
Change in clinical signs of rostral displacement of fluids | 28 days
Tolerance overall judgment and questionnaire and adverse events) | 28 days (only during the phase with the wearing of compression stockings
  overall judgment by the patient and questionnaire filled by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Pathologies du Sommeil Bâtiment EOLE GH Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No